CLINICAL TRIAL: NCT00089544
Title: A Pilot Phase II Study of Pre-Operative Radiation Therapy and Thalidomide (IND 48832; NSC 66847) for Low Grade Primary Soft Tissue Sarcoma or Pre-Operative MAID/Thalidomide/Radiation Therapy for High/Intermediate Grade Primary Soft Tissue Sarcoma of the Extremity or Body Wall
Brief Title: Preoperative Thalidomide With Radiation Therapy For Patients With Low-Grade Primary Soft Tissue Sarcoma or Thalidomide With Radiation Therapy and Chemotherapy For Patients With High-Grade or Intermediate-Grade Primary Soft Tissue Sarcoma of the Arm, Leg, or Body Wall
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02588; NCI-2012-02588 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RTOG-0330; CDR0000365499; RTOG-0330 (Other: Radiation Therapy Oncology Group); RTOG-0330 (Other: CTEP); U10CA021661 (NIH)
Record Dates: First submitted 2004-08-06; First posted 2004-08-09 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-03

CONDITIONS: Recurrent Adult Soft Tissue Sarcoma; Stage I Adult Soft Tissue Sarcoma AJCC v7; Stage II Adult Soft Tissue Sarcoma AJCC v7; Stage III Adult Soft Tissue Sarcoma AJCC v7
MeSH Terms: conditions — Sarcoma | interventions — Dacarbazine; Doxorubicin; Filgrastim; Granulocyte Colony-Stimulating Factor; Ifosfamide; Radiotherapy; Radiation; Thalidomide

ARMS (2):
- Cohort A (chemotherapy, radiation, thalidomide, surgery) (Experimental): Patients receive doxorubicin, ifosfamide, and dacarbazine IV continuously on days 1-3, 22-24, and 43-45. Patients receive G-CSF subcutaneously beginning on days 4, 25, and 46 and continuing until blood counts recover. Patients undergo radiotherapy once daily on days 7-11, 14-18, 21, 28-32, 35-39, and 42. Patients receive oral thalidomide once daily on days 7-21 and 26-42. Patients undergo surgical resection between days 84 and 98. Beginning 2 weeks after surgery, patients receive oral thalidomide once daily for 12 months in the absence of unacceptable toxicity.
  Interventions: Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Biological: Filgrastim; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Radiation: Radiation Therapy; Drug: Thalidomide; Procedure: Therapeutic Conventional Surgery
- Cohort B (thalidomide, radiation, surgery) (Experimental): Patients receive oral thalidomide once daily beginning on day 1 and continuing until 1 week before surgery. Patients undergo radiotherapy once daily, 5 days a week, on weeks 1-5. Patients undergo surgical resection between days 77 and 91. Beginning 2 weeks after surgery, patients receive oral thalidomide once daily for 6 months in the absence of unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Radiation: Radiation Therapy; Drug: Thalidomide; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
  Arms: Cohort A (chemotherapy, radiation, thalidomide, surgery)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
  Arms: Cohort A (chemotherapy, radiation, thalidomide, surgery)
Biological: Filgrastim — Given subcutaneously
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
  Arms: Cohort A (chemotherapy, radiation, thalidomide, surgery)
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
  Arms: Cohort A (chemotherapy, radiation, thalidomide, surgery)
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Radiation Therapy — Undergo radiotherapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; RADIATION; Radiotherapeutics; radiotherapy; RT; Therapy, Radiation
Drug: Thalidomide — Given orally
  Other Names: (+)-Thalidomide; (-)-Thalidomide; .alpha.-Phthalimidoglutarimide; 2, 6-Dioxo-3-phthalimidopiperidine; Alpha-Phthalimidoglutarimide; Contergan; Distaval; Kevadon; N-(2,6-Dioxo-3-piperidyl)phthalimide; N-Phthaloylglutamimide; N-Phthalylglutamic Acid Imide; Neurosedyn; Pantosediv; Phthalimide, N-(2, 6-dioxo-3-piperidyl)-, (+)-; Phthalimide, N-(2, 6-dioxo-3-piperidyl)-, (-)-; Sedalis; Sedoval K-17; Softenon; Synovir; Talimol; Thalomid
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection

SUMMARY:
Thalidomide may stop the growth of soft tissue sarcoma by stopping blood flow to the tumor. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy, such as doxorubicin, ifosfamide, and dacarbazine, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving thalidomide together with radiation therapy and/or chemotherapy before surgery may shrink the tumor so that it can be removed. This phase II trial is studying how well giving preoperative (before surgery) thalidomide together with radiation therapy works in treating patients with low-grade primary soft tissue sarcoma, and how well giving thalidomide together with radiation therapy, doxorubicin, ifosfamide, and dacarbazine works in treating patients with high-grade or intermediate-grade primary soft tissue sarcoma of the arm, leg, chest wall, or abdominal wall.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the treatment delivery and toxicity of the combination of thalidomide and radiotherapy in patients with low-grade primary soft tissue sarcoma of the extremity or body wall.

II. Determine the treatment delivery and toxicity of the combination of thalidomide and doxorubicin, ifosfamide, dacarbazine, and radiotherapy in patients with high- or intermediate-grade primary soft tissue sarcoma of the extremity or body wall and compare these results with those of patients treated on RTOG-9514.

III. Determine the feasibility of using specific tissue and circulating biomarkers of antiangiogenic response in patients treated with these regimens, in a multi-institutional setting.

IV. Determine the quantitative changes and patient variabilities of these biomarkers before, during, and after therapy with these regimens.

V. Determine the baseline data sets of biomarkers, particularly circulating endothelial cells, in patients treated with these regimens.

VI. Determine the tolerance to long-term post-operative thalidomide in these patients.

VII. Determine the clinical response to pre-operative therapy in these patients.

VIII. Correlate local control and disease-free survival with surrogate biological endpoints in patients treated with these regimens.

OUTLINE: This is a pilot, cohort study. Patients with high- or intermediate-grade tumors >= 8 cm in diameter are assigned to cohort A and patients with low-grade tumors > 5 cm in diameter are assigned to cohort B.

Cohort A: Patients receive doxorubicin, ifosfamide, and dacarbazine IV continuously on days 1-3, 22-24, and 43-45. Patients receive filgrastim (G-CSF) subcutaneously beginning on days 4, 25, and 46 and continuing until blood counts recover. Patients undergo radiotherapy once daily on days 7-11, 14-18, 21, 28-32, 35-39, and 42. Patients receive oral thalidomide once daily on days 7-21 and 26-42. Patients undergo surgical resection between days 84 and 98. Beginning 2 weeks after surgery, patients receive oral thalidomide once daily for 12 months in the absence of unacceptable toxicity.

Cohort B: Patients receive oral thalidomide once daily beginning on day 1 and continuing until 1 week before surgery. Patients undergo radiotherapy once daily, 5 days a week, on weeks 1-5. Patients undergo surgical resection between days 77 and 91. Beginning 2 weeks after surgery, patients receive oral thalidomide once daily for 6 months in the absence of unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 44 patients (22 per cohort) will be accrued for this study within 17 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary soft tissue sarcoma

  * T2a or T2b disease
  * Superficial or deep tumor
  * Grade 1, 2, 3, or 4
  * Tumor located on the upper extremity (including shoulder), lower extremity (including hip), or trunk
* Meets 1 of the following criteria:

  * Tumor ? 8 cm in maximal diameter and grade 3 or 4 (intermediate or high grade) (cohort A)
  * Tumor > 5 cm in maximal diameter and grade 1 or 2 (low grade) (cohort B)
* Locally recurrent disease allowed provided there has been no prior radiotherapy to the primary tumor
* No histologically confirmed rhabdomyosarcoma, extraosseous Ewing's primitive neuroectodermal tumors, osteosarcoma or chondrosarcoma, Kaposi's sarcoma, angiosarcoma, desmoid tumors, or dermatofibrosarcoma protuberans
* No overt evidence of lung metastases (CT scan evidence of small incidental lesions without histologic diagnosis allowed)
* No evidence of other metastases
* No sarcoma of the head, neck, intra-abdominal, or retroperitoneal region
* Performance status - Zubrod 0-1
* At least 2 years
* Absolute neutrophil count ? 1,500/mm^3
* Platelet count ? 120,000/mm^3
* Hemoglobin ? 8.0 g/dL (cohort A)
* No known hypercoagulable disorders, such as the following:

  * APC resistance (factor V Leiden)
  * Protein S deficiency
  * Protein C deficiency
  * Antithrombin III deficiency
  * Hyperhomocystinemia
  * Dysplasminogenemia
  * High plasminogen activator inhibitor
  * Dysfibrinogenemia
  * Antiphospholipid syndrome
  * Thrombocythemia
  * Dysproteinemia
* Fibrin split products < 2 times upper limit of normal (ULN)
* Fibrinogen > 200 mg/dL
* Bilirubin ? 1.5 mg/dL (1.0 mg/dL for patients with Gilbert's syndrome)
* AST and ALT ? 2.0 times ULN
* PT and PTT < 1.25 times ULN (except in patients treated with anticoagulants for unrelated medical conditions [e.g., atrial fibrillation])
* No history of hepatic cirrhosis
* Creatinine ? 1.5 mg/dL
* Creatinine clearance > 60 mL/min
* No atherosclerotic coronary artery disease that required bypass surgery within the past year
* No uncompensated coronary artery disease by ECG or physical examination
* No myocardial infarction within the past 6 months
* No severe or unstable angina within the past 6 months
* No uncompensated congestive heart failure
* No New York Heart Association class II-IV heart disease
* No symptomatic peripheral vascular disease
* No history of deep vein thrombosis
* Cohort A only:

  * EF ? 50% within the past 6 months
  * LVEF > 50%
* No pulmonary embolus except if caused directly by foreign body implants (e.g., central venous catheters or portacaths)
* No global neurocognitive symptomatology
* No fatigue ? grade 2
* No history of uncontrolled seizures or uncontrolled seizure disorder
* No sensory neuropathy ? grade 2 except for localized neuropathy due to mechanical cause or trauma
* No other malignancies within the past 3 years except non-invasive malignancies (e.g., carcinoma in situ of the cervix, breast, or oral cavity) or squamous or basal cell skin cancer
* No history of uncontrolled myxedema
* No hypothyroidism ? grade 3
* No active uncontrolled bacterial, viral, or fungal infection
* No other significant illness that would preclude surgery
* No other major illness or psychiatric impairment that would preclude study therapy
* No known AIDS
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective barrier methods of contraception for 4 weeks before, during, and for at least 4 weeks after study treatment
* No prior thalidomide
* No prior biologic therapy for this tumor
* No prior chemotherapy for this tumor
* See Disease Characteristics
* No prior radiotherapy for this tumor
* See Cardiovascular
* No other concurrent investigational drugs
* No concurrent sedating drugs
* No concurrent illegal sedating "recreational" drugs
* No concurrent alcohol intake of more than 1 drink per day

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-06-17 (Actual); Primary Completion 2011-09-27 (Actual); Study Completion 2013-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burton Eisenberg, Principal Investigator — Radiation Therapy Oncology Group
Locations (1):
- Radiation Therapy Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (Chemotherapy, Radiation, Thalidomide, Surgery): Patients receive doxorubicin, ifosfamide, and dacarbazine IV continuously on days 1-3, 22-24, and 43-45. Patients receive G-CSF subcutaneously beginning on days 4, 25, and 46 and continuing until blood counts recover. Patients undergo radiotherapy once daily on days 7-11, 14-18, 21, 28-32, 35-39, and 42. Patients receive oral thalidomide once daily on days 7-21 and 28-42. Patients undergo surgical resection between days 84 and 98. Beginning 2 weeks after surgery, patients receive oral thalidomide once daily for 12 months in the absence of unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort A (Chemotherapy, Radiation, Thalidomide, Surgery) | Cohort B (Thalidomide, Radiation, Surgery)
Started | 16 | 7
Completed | 15 (Subjects contributing data to the primary analysis are considered to have completed the study.) | 7
Not Completed | 1 | 0
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients who started treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Chemotherapy, Radiation, Thalidomide, Surgery) | Cohort B (Thalidomide, Radiation, Surgery) | Total
Number analyzed (Participants) | 15 | 7 | 22
Age, Continuous [Median (Full Range); unit: years] | 49.0 [20.0 to 75.0] | 47.0 [39.0 to 81.0] | 48 [20 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Treatment Delivery With Compliance Defined as Receiving at Least 95% of the Pre-operative Protocol Dose of RT, All 3 Cycles of MAID (if Applicable), and Receive Thalidomide on 75% of the Days During Radiation
Description: Was to be estimated using a binomial distribution and accompanied by the associated 95% confidence interval. Due to early study closure, this endpoint could not be fully evaluated per the protocol plan.
Time Frame: Duration of treatment (which can continue up to approximately 15 months).
Population: Eligible patients who started study treatment.
Measure: Number; unit: participants
Arm/Group | Cohort A (Chemotherapy, Radiation, Thalidomide, Surgery) | Cohort B (Thalidomide, Radiation, Surgery)
Number analyzed (Participants) | 15 | 7
participants
  Not Compliant | 5 | 2
  Compliant | 10 | 5

2. Secondary Outcome: Wound Complication (Grades 2, 3, 4, and 5) as Measured by CTCAE v3.0
Description: Will be estimated using a binomial distribution and accompanied by the associated 95% confidence interval.
Time Frame: From start of treatment to time of surgery
Population: This analysis was not carried out due to the small number of patients accrued to the study. See section "Limitations and Caveats".
Arm/Group | Cohort A (Chemotherapy, Radiation, Thalidomide, Surgery) | Cohort B (Thalidomide, Radiation, Surgery)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Response to Pre-operative Therapy Assessed Using RECIST Criteria
Time Frame: From start of treatment to time of surgery.
Population: as for outcome 2
Arm/Group | Cohort A (Chemotherapy, Radiation, Thalidomide, Surgery) | Cohort B (Thalidomide, Radiation, Surgery)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Per the protocol, toxicity data was collected via CTCAE3.0 then mapped to CTCAE 4.0 for reporting on this website. Subjects experiencing more than one of a given SAE are counted only once for that SAE. Subjects experiencing more than one of a given "Other (Not Including Serious)" AE are counted only once for that "Other (Not Including Serious)" AE.
Arm/Group | Cohort A (Chemotherapy, Radiation, Thalidomide, Surgery) | Cohort B (Thalidomide, Radiation, Surgery)
Serious Adverse Events (participants affected / at risk) | 9/15 | 3/7
Other Adverse Events (participants affected / at risk) | 15/15 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Chemotherapy, Radiation, Thalidomide, Surgery) (N=15) | Cohort B (Thalidomide, Radiation, Surgery) (N=7)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Edema limbs (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 4 | 0
Platelet count decreased (Investigations) | 3 | 0
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 5 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 5 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Chemotherapy, Radiation, Thalidomide, Surgery) (N=15) | Cohort B (Thalidomide, Radiation, Surgery) (N=7)
Anemia (Blood and lymphatic system disorders) | 13 | 2
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 4 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Blurred vision (Eye disorders) | 3 | 0
Extraocular muscle paresis (Eye disorders) | 0 | 1
Watering eyes (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal hemorrhage (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 11 | 3
Diarrhea (Gastrointestinal disorders) | 4 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 13 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 10 | 0
Edema limbs (General disorders) | 6 | 1
Fatigue (General disorders) | 14 | 4
Fever (General disorders) | 5 | 0
Gait disturbance (General disorders) | 2 | 0
Hypothermia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 0
Allergic reaction (Immune system disorders) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 2 | 0
Joint infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 5 | 3
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 | 1
Seroma (Injury, poisoning and procedural complications) | 2 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 3 | 2
Alanine aminotransferase increased (Investigations) | 5 | 0
Alkaline phosphatase increased (Investigations) | 6 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood bilirubin increased (Investigations) | 3 | 0
Creatinine increased (Investigations) | 2 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0
Haptoglobin decreased (Investigations) | 1 | 0
INR increased (Investigations) | 0 | 1
Investigations - Other (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 5 | 0
Neutrophil count decreased (Investigations) | 6 | 0
Platelet count decreased (Investigations) | 3 | 0
Weight loss (Investigations) | 3 | 0
White blood cell decreased (Investigations) | 8 | 0
Anorexia (Metabolism and nutrition disorders) | 8 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 6 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 0
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 0
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 3 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 3
Phantom pain (Nervous system disorders) | 1 | 0
Sinus pain (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Confusion (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 2 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 4 | 0
Thromboembolic event (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study closed early due to unacceptably high rate of thromboembolic events in Cohort A and due to low accrual in Cohort B. For this reason efficacy endpoints other than response to pre-operative therapy were not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less